CLINICAL TRIAL: NCT03984604
Title: A Double-Blind, Randomized, Placebo-Controlled, Multi-Center Dose-Titration Study on the Efficacy and Safety of CHI-921 on Sleep Initiation and Maintenance in Subjects With Insomnia
Brief Title: Investigation of the Efficacy and Safety of CHI-921 in Insomnia.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Canopy Growth Corporation (Industry)
Collaborators: Galenova Inc (Other); Algorithme Pharma Inc (Industry); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2017-01
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2019-08

CONDITIONS: Insomnia
Keywords: sleep; cannabis; primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHI-921 (Active Comparator): During the double-blind treatment period (9 weeks), subjects will take 0.5 mL of their randomized treatment (CHI-921) for 3 weeks, followed by another 3 weeks of treatment at 1.0 mL for and another 3 weeks of treatment at 2.0 mL.
  Interventions: Drug: CHI-921
- Placebo (Placebo Comparator): During the double-blind treatment period (9 weeks), subjects will take 0.5 mL of their randomized treatment (placebo) for 3 weeks, followed by another 3 weeks of placebo treatment at 1.0 mL for and another 3 weeks of placebo treatment at 2.0 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHI-921 — a standardized cannabis extract in sunflower oil administered in oral liquid (oil) form
  Arms: CHI-921
Drug: Placebo — Placebo is a vehicle oil will match CHI-921
  Arms: Placebo

SUMMARY:
Insomnia is a disorder where people are having trouble sleeping and can include difficulty falling asleep, staying asleep and waking up too early, as well as having unrefreshing sleep. CHI-921 is a cannabis extract in sunflower oil produced as a treatment for insomnia. This trial is designed to evaluate the efficacy and safety of CHI-921 on people with insomnia.

DETAILED DESCRIPTION:
The study is designed to:

1. Evaluate the patient-reported sleep latency and patient-reported wake after sleep onset after 3 weeks per treatment dose with CHI-921 compared to placebo.
2. To evaluate the effects of CHI-921 compared to placebo on PSG sleep architecture.
3. To evaluate the effects of CHI-921 compared to placebo on Patient Global Impression of change.
4. To evaluate the daytime residual effects that may be associated with CHI-921 as compared to placebo during the double-blind treatment period using patient's morning and evening questionnaire, Clinical Global Impression of change, Insomnia Severity Index, Pittsburgh Sleep Quality Index, Epworth Sleepiness Scale as well as the Rey Auditory Verbal Learning Test and Digit Symbol Substitution psychometric tests.
5. To assess the effect on sleep of abruptly discontinuing CHI-921 compared to placebo (during run-out period).
6. To evaluate the clinical safety and tolerability of CHI-921 compared to placebo.
7. Evaluation of the accuracy of sleep data obtained by actigraphy as compared to traditional PSG.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects 25 to 70 years of age, inclusive
2. Willing and able to give informed consent for study participation
3. Each patient must have insomnia disorder based on criteria (ICSD-3 or DSM-5) with predominant complaints of difficulty in initiating or maintaining sleep for at least three months preceding the study visit and having clinically significant distress or impairment in social occupational or other important areas of functioning
4. Normal vital signs as follows:

   * Sitting systolic blood pressure (SBP) between 90 and 140 mmHg, inclusive
   * Sitting diastolic blood pressure (DBP) between 55 and 90 mmHg, inclusive
   * Pulse rate between 50 and 100 bpm inclusive
5. Willing to comply with all study requirements and procedures for the duration of the clinical study
6. Willing to comply with the study restrictions including:

   * Adherence to concomitant drug washout requirements, as applicable, for the duration of the clinical study
   * Willing to abstain from alcohol for the duration of the clinical study
   * Willing to abstain from caffeine 10 hours before each recording
   * If a smoker, willing to abstain from smoking at night from approximately 10 pm to 8 am for the duration of the clinical study
7. Female subjects who:

   * Are postmenopausal, with amenorrhea for at least 1 year before the screening visit,
   * Are surgically sterile, OR
   * If of childbearing potential agree to practice effective double barrier methods of contraception, from the time of the signing of informed consent through the last dose of study drug and for 30 days after dosing stops (1 ovulatory cycle), or agree to completely abstain from intercourse
   * Males with female partners of childbearing potential are also expected to practice effective barrier methods of contraception from the time of signing informed consent through the last dose of study drug and for 30 days after dosing stops.
8. Self-reported bedtime between 9 pm and midnight on 4-7 nights per week
9. Based on the PSG recordings during the screening nights (V2; SN1 and SN2), one of the following criteria must be present:

   1. Mean WASO calculated on SN1 and SN2 > 30 min or
   2. Mean LPS: calculated on SN1 and SN2 > 30 min

Exclusion Criteria

1. Body mass index > 32 calculated from patient's height (m) and weight (kg); weight (kg)/square height (m²)
2. Presence of a sleep disorder (for sleep apnea syndrome, an apnea-hypopnea index > 15 per hour of sleep on the first screening night will be used as an exclusion criterion; for periodic limb movement disorder, an index of periodic limb movements during sleep associated with an arousal > 10 per hour of sleep on the first screening night will be used as an exclusion criterion)
3. Patients with a history of epilepsy or seizures (not including benign neonatal and childhood convulsions)
4. Serious head injury or stroke within the past year
5. Any evidence of psychiatric disorder (including Beck Depression Inventory [BDI] ≥ 20) and/or history of psychosis excluding insomnia
6. Evidence of any clinically significant, severe or unstable, acute or chronically progressive medical or surgical disorder (including planned medical procedures that may impact sleep), or any condition that may interfere with the absorption, metabolism, distribution, or excretion of the study drug, or may affect patient safety
7. Clinically significant and abnormal electrocardiogram (ECG; including QTc ≥ 450 ms for males, 460 ms for females) or patients with a history of cardiovascular disease including poorly controlled hypertension, ischaemic heart disease, arrhythmia, or severe heart failure
8. Positive qualitative urine drug screen (opiates, cocaine, amphetamine, cannabinoids, barbiturates, phencyclidine, benzodiazepines, methadone, propoxyphene), at screening
9. Use of any substance with psychotropic effects or properties known to affect sleep/wake, including neuroleptics, morphine/opioid derivatives, antihistamines, stimulants antidepressants, clonidine, within one week or five half-lives (whichever is longer) prior to screening
10. Use of any over-the-counter sleep medications including tryptophan, valerian root (Valeriana officinalis), kava (Piper methysticum Forst), melatonin, St John's Wort (Hypericum perforatum), Alluna (herbal sleep supplement with valerian root), and hemp within 1 week or 5 half-lives (whichever is longer) prior to screening
11. Consumption of xanthine-containing beverages (i.e., tea, coffee, or cola) of more than 5 cups or glasses per day
12. Participation in any other trial within 30 days before the screening visit
13. Night shift workers (during the 12 months prior to the study and during the study)
14. Individuals who nap 3 or more times per week over the preceding month
15. Individuals having to travel across more than 3 time zones in the month prior to screening or individuals who plan on travelling outside of their country of residence at any time during the study
16. Other exclusion criteria based on adverse events (AE) or serious adverse events (SAE) reported in the Investigator Brochure
17. Women who are pregnant, are planning to become pregnant, or are breastfeeding
18. Individuals may be excluded from participating in the study based on the investigator's professional judgement

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline of PSG latency to persistent sleep | after 3 weeks per treatment dose with CHI-921 compared to placebo
Change from baseline of PSG wake after sleep onset (WASO) | after 3 weeks per treatment dose with CHI-921 compared to placebo

SECONDARY OUTCOMES:
Change from baseline of patient-reported mean sleep latency (subjective sleep latency). | after 3 weeks of treatment
Change from baseline of patient-reported mean wake after sleep onset (subjective WASO) | after 3 weeks of treatment
Change from baseline on PSG sleep architecture: percentage of total sleep spent in each sleep stage (N1, N2, N3 and rapid eye movement [REM] sleep) | after 3 weeks of treatment
Patient Global Impression of change (PGI-c) | Visit 2/Screening Night 1, Visit 4/Night 21, Visit 5/Night 42, Visit 6/Night 63
  Standard 7 question index
Clinical Global Impression of change (CGI-c) | Visit 2/Screening Night 1, Visit 4/Night 21, Visit 5/Night 42, Visit 6/Night 63
  Standard 7 question index
Insomnia Severity Index (ISI) | Visit 2/Screening Night 1, Visit 4/Night 21, Visit 5/Night 42, Visit 6/Night 63
  Standard 7 question index
Pittsburgh Sleep Quality Index (PSQI) | Visit 2/Screening Night 1, Visit 4/Night 21, Visit 5/Night 42, Visit 6/Night 63
  Standard 10 question index
Epworth Sleepiness Scale (ESS) | Visit 2/Screening Night 1, Visit 4/Night 21, Visit 5/Night 42, Visit 6/Night 63
  Standard 8 question index
Rey Auditory Verbal Learning Test | Visit 2/Screening Night 1 and 2, Visit 3/ Night 1, Visit 4/Night 21 and 22, Visit 5/Night 42 and 43, Visit 6/Night 63
Digit Symbol Substitution Test | Visit 2/Screening Night 1 and 2, Visit 3/ Night 1, Visit 4/Night 21 and 22, Visit 5/Night 42 and 43, Visit 6/Night 63

CONTACTS AND LOCATIONS:
Overall Officials: Dr M Ware, MD, Study Director — Canopy Growth Corporation
Locations (1):
- Algorithme Pharma Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No